CLINICAL TRIAL: NCT03436472
Title: Impact of Dexmedetomidine on Long-term Outcome in Elderly Patients After Noncardiac Surgery: 5-year Follow-up of a Randomized Controlled Trial
Brief Title: Dexmedetomidine and 5-year Outcome in Elderly Patients After Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Peking University First Hospital (Other)
Collaborators: Peking University Third Hospital (Other)
Responsible Party: Principal Investigator, Dong-Xin Wang, Professor and Chairman, Department of Anesthesiology and Critical Care Medicine, Peking University First Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: Dex-5-2016
Record Dates: First submitted 2018-02-12; First posted 2018-02-19 (Actual); Last update posted 2019-06-21 (Actual); Status verified 2019-06

CONDITIONS: Aged; Operative; Delirium; Dexmedetomidine; Mortality; Long-term Survivors
Keywords: aged; operative; delirium; dexmedetomidine; long-term outcome
MeSH Terms: conditions — Delirium | interventions — Dexmedetomidine; Saline Solution; Sodium Chloride

STUDY DESIGN:
Intervention Model Description: Parallel Assignment
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- dexmedetomidine group (Experimental): For patients who were not intubated, dexmedetomidine was infused at a rate of 0.1 microgram/kg per hour from study recruitment on the day of surgery until 8:00 am on the first day after surgery. For patients who were intubated and mechanically ventilated, dexmedetomidine infusion was started after the Richmond Agitation Sedation Scale was -2 or higher after intensive care unit admission until 8:00 am on the first day after surgery.
  Interventions: Drug: dexmedetomidine
- placebo group (Placebo Comparator): Normal saline was infused in the same rate for the same duration as that in the placebo group.
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: dexmedetomidine — low-dose dexmedetomidine infusion
  Other Names: dexmedetomidine hydrochloride
  Arms: dexmedetomidine group
Drug: placebo — normal saline infusion
  Other Names: normal saline; 0.9% sodium chloride
  Arms: placebo group

SUMMARY:
Delirium is a frequent postoperative complication. Its occurrence is associated with worse long-term outcomes. In a previous randomized controlled trial, prophylactic low-dose dexmedetomidine infusion during the early postoperative period decreased the incidence of delirium in elderly patients after surgery. The purpose of this 5-year follow-up study is to evaluate whether prophylactic low-dose dexmedetomidine infusion can improve the 5-year outcomes in elderly patients recruited in the previous randomized controlled trial.

DETAILED DESCRIPTION:
Delirium is a frequent postoperative complication; a systematic review revealed that postoperative delirium occurs in 36.8% of surgical patients, and its prevalence increases with age. The occurrence of delirium is associated with worse long-term outcomes including worse functional recovery, decline in cognitive function, and increased mortality rate. Surgical stress, pain, and sleep disturbances are important factors leading to postoperative delirium in the elderly.

Dexmedetomidine is a highly selective alpha-2 adrenoreceptor agonist that provides anti-anxiety, sedation, and modest analgesia with minimal respiratory depression. For mechanically ventilated intensive care unit (ICU) patients, dexmedetomidine sedation improves the quality of sleep, decreases the incidence of delirium, and shortens the duration of ICU stay. For patients undergoing surgery, perioperative dexmedetomidine relieves the severity of stress response, decreases the requirement of anesthetics, and improves postoperative analgesia.

In the previous stage of the current study, 700 elderly patients who were admitted to the ICU after noncardiac surgery were recruited and randomized into two groups (dexmedetomidine group and placebo [normal saline] group). The results showed that prophylactic low-dose dexmedetomidine infusion during the early postoperative period ameliorated the subjective sleep quality and decreased the incidence of delirium (22.6% [79/350] with placebo vs. 9.1% [32/350] with dexmedetomidine; odds ratio 0.35, 95% confidence interval 0.22 to 0.54; p < 0.0001). The investigators hypothesize that low-dose dexmedetomidine infusion may also improve long-term outcome in this patient population.

The purpose of this 5-year follow-up study is to evaluate whether prophylactic low-dose dexmedetomidine infusion during the early postoperative period can improve the 5-year outcomes in elderly patients recruited in the previous randomized controlled trial.

ELIGIBILITY:
Inclusion Criteria:

Patients were included if they met all of the following criteria:

* Age of 65 years or older;
* Underwent elective noncardiac surgery under general anesthesia;
* Admitted to ICU after surgery.

Exclusion Criteria:

Patients were excluded if they met any of the following criteria:

* Preoperative history of schizophrenia, epilepsy, Parkinsonism or myasthenia gravis;
* Inability to communicate in the preoperative period (because of coma, profound dementia or language barrier);
* Brain injury or neurosurgery;
* Preoperative left ventricular ejection fraction < 30%, sick sinus syndrome, severe sinus bradycardia (< 50 beats per minute), or second-degree or greater atrioventricular block without pacemaker;
* Serious hepatic dysfunction (Child-Pugh class C);
* Serious renal dysfunction (undergoing dialysis before surgery); or
* Unlikely to survive for more than 24 hours.

Ages: 65 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Gender Based: Yes
Enrollment: 700 (Actual)
Dates: Start 2017-06-01 (Actual); Primary Completion 2019-01-08 (Actual); Study Completion 2019-04-01 (Actual)

PRIMARY OUTCOMES:
Duration of 5-year survival after surgery | From the day of surgery until the end of the 5th year after surgery
  Duration of 5-year survival after surgery

SECONDARY OUTCOMES:
Survival rates after surgery | At 6 months, 1 year, 2 years ,3 years, 4 years,and 5 years after surgery
  Survival rates at different timepoints after surgery
Cognitive function in 5-year survivors after surgery | At the end of the 5th year after surgery
  Cognitive function is assessed with Telephone Interview for Cognitive Status-Modified (TICS-M).
Health related quality of life in 5-year survivors after surgery | At the end of the 5th year after surgery
  Health related quality of life is assessed with World Health Organization Quality of Life-BREF (WHOQOL-BREF).

OTHER OUTCOMES:
Survival rates in the subgroup of patients after cancer or non-cancer surgery | At 6 months, 1 year, 2 years, 3 years, 4 years, and 5 years after surgery
  Survival rates at different time-points in the subgroup of patients after cancer or non-cancer surgery
Duration of survival in the subgroup of patients after cancer or non-cancer surgery | From the day of surgery until the end of the 5th year after surgery
  Duration of survival in the subgroup of patients after cancer or non-cancer surgery
Cognitive function in the subgroup of 5-year survivors after cancer or non-cancer surgery | At the end of the 5th year after surgery
  Cognitive function is assessed with Telephone Interview for Cognitive Status-Modified (TICS-M)
Health related quality of life in the subgroup of 5-year survivors after cancer or non-cancer surgery | At the end of the 5th year after surgery
  Health related quality of life is assessed with World Health Organization Quality of Life-BREF (WHOQOL-BREF).

CONTACTS AND LOCATIONS:
Overall Officials: Dong-Xin Wang, MD,PhD, Principal Investigator — Peking University First Hospital
Locations (1):
- Peking University First Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: No
Data will be provided on request.

REFERENCES:
- [Background] Rabe-Jablonska J, Bienkiewicz W. [Anxiety disorders in the fourth edition of the classification of mental disorders prepared by the American Psychiatric Association: diagnostic and statistical manual of mental disorders (DMS-IV -- options book]. Psychiatr Pol. 1994 Mar-Apr;28(2):255-68. Polish. PMID 8208869
- [Background] Dyer CB, Ashton CM, Teasdale TA. Postoperative delirium. A review of 80 primary data-collection studies. Arch Intern Med. 1995 Mar 13;155(5):461-5. doi: 10.1001/archinte.155.5.461. PMID 7864702
- [Background] Girard TD, Pandharipande PP, Ely EW. Delirium in the intensive care unit. Crit Care. 2008;12 Suppl 3(Suppl 3):S3. doi: 10.1186/cc6149. Epub 2008 May 14. PMID 18495054
- [Background] Mu DL, Wang DX, Li LH, Shan GJ, Li J, Yu QJ, Shi CX. High serum cortisol level is associated with increased risk of delirium after coronary artery bypass graft surgery: a prospective cohort study. Crit Care. 2010;14(6):R238. doi: 10.1186/cc9393. Epub 2010 Dec 30. PMID 21192800
- [Background] Shi CM, Wang DX, Chen KS, Gu XE. Incidence and risk factors of delirium in critically ill patients after non-cardiac surgery. Chin Med J (Engl). 2010 Apr 20;123(8):993-9. PMID 20497703
- [Background] Roberts B, Rickard CM, Rajbhandari D, Turner G, Clarke J, Hill D, Tauschke C, Chaboyer W, Parsons R. Multicentre study of delirium in ICU patients using a simple screening tool. Aust Crit Care. 2005 Feb;18(1):6, 8-9, 11-4 passim. doi: 10.1016/s1036-7314(05)80019-0. PMID 18038529
- [Background] Balas MC, Happ MB, Yang W, Chelluri L, Richmond T. Outcomes Associated With Delirium in Older Patients in Surgical ICUs. Chest. 2009 Jan;135(1):18-25. doi: 10.1378/chest.08-1456. Epub 2008 Nov 18. PMID 19017895
- [Background] Ely EW, Gautam S, Margolin R, Francis J, May L, Speroff T, Truman B, Dittus R, Bernard R, Inouye SK. The impact of delirium in the intensive care unit on hospital length of stay. Intensive Care Med. 2001 Dec;27(12):1892-900. doi: 10.1007/s00134-001-1132-2. Epub 2001 Nov 8. PMID 11797025
- [Background] Ansaloni L, Catena F, Chattat R, Fortuna D, Franceschi C, Mascitti P, Melotti RM. Risk factors and incidence of postoperative delirium in elderly patients after elective and emergency surgery. Br J Surg. 2010 Feb;97(2):273-80. doi: 10.1002/bjs.6843. PMID 20069607
- [Background] Ely EW, Shintani A, Truman B, Speroff T, Gordon SM, Harrell FE Jr, Inouye SK, Bernard GR, Dittus RS. Delirium as a predictor of mortality in mechanically ventilated patients in the intensive care unit. JAMA. 2004 Apr 14;291(14):1753-62. doi: 10.1001/jama.291.14.1753. PMID 15082703
- [Background] Franco K, Litaker D, Locala J, Bronson D. The cost of delirium in the surgical patient. Psychosomatics. 2001 Jan-Feb;42(1):68-73. doi: 10.1176/appi.psy.42.1.68. PMID 11161124
- [Background] Milbrandt EB, Deppen S, Harrison PL, Shintani AK, Speroff T, Stiles RA, Truman B, Bernard GR, Dittus RS, Ely EW. Costs associated with delirium in mechanically ventilated patients. Crit Care Med. 2004 Apr;32(4):955-62. doi: 10.1097/01.ccm.0000119429.16055.92. PMID 15071384
- [Background] Pisani MA, Kong SY, Kasl SV, Murphy TE, Araujo KL, Van Ness PH. Days of delirium are associated with 1-year mortality in an older intensive care unit population. Am J Respir Crit Care Med. 2009 Dec 1;180(11):1092-7. doi: 10.1164/rccm.200904-0537OC. Epub 2009 Sep 10. PMID 19745202
- [Background] Bickel H, Gradinger R, Kochs E, Forstl H. High risk of cognitive and functional decline after postoperative delirium. A three-year prospective study. Dement Geriatr Cogn Disord. 2008;26(1):26-31. doi: 10.1159/000140804. Epub 2008 Jun 24. PMID 18577850
- [Background] Van Rompaey B, Schuurmans MJ, Shortridge-Baggett LM, Truijen S, Elseviers M, Bossaert L. Long term outcome after delirium in the intensive care unit. J Clin Nurs. 2009 Dec;18(23):3349-57. doi: 10.1111/j.1365-2702.2009.02933.x. Epub 2009 Sep 4. PMID 19735334
- [Background] Vaurio LE, Sands LP, Wang Y, Mullen EA, Leung JM. Postoperative delirium: the importance of pain and pain management. Anesth Analg. 2006 Apr;102(4):1267-73. doi: 10.1213/01.ane.0000199156.59226.af. PMID 16551935
- [Background] Halaszynski TM. Pain management in the elderly and cognitively impaired patient: the role of regional anesthesia and analgesia. Curr Opin Anaesthesiol. 2009 Oct;22(5):594-9. doi: 10.1097/ACO.0b013e32833020dc. PMID 19623056
- [Background] Hudek K. Emergence delirium: a nursing perspective. AORN J. 2009 Mar;89(3):509-16; quiz 517-9. doi: 10.1016/j.aorn.2008.12.026. PMID 19326585
- [Background] Rudolph JL, Ramlawi B, Kuchel GA, McElhaney JE, Xie D, Sellke FW, Khabbaz K, Levkoff SE, Marcantonio ER. Chemokines are associated with delirium after cardiac surgery. J Gerontol A Biol Sci Med Sci. 2008 Feb;63(2):184-9. doi: 10.1093/gerona/63.2.184. PMID 18314455
- [Background] de Rooij SE, van Munster BC, Korevaar JC, Levi M. Cytokines and acute phase response in delirium. J Psychosom Res. 2007 May;62(5):521-5. doi: 10.1016/j.jpsychores.2006.11.013. PMID 17467406
- [Background] Roth-Isigkeit A, Borstel TV, Seyfarth M, Schmucker P. Perioperative serum levels of tumour-necrosis-factor alpha (TNF-alpha), IL-1 beta, IL-6, IL-10 and soluble IL-2 receptor in patients undergoing cardiac surgery with cardiopulmonary bypass without and with correction for haemodilution. Clin Exp Immunol. 1999 Nov;118(2):242-6. doi: 10.1046/j.1365-2249.1999.01050.x. PMID 10540185
- [Background] Holmes JH 4th, Connolly NC, Paull DL, Hill ME, Guyton SW, Ziegler SF, Hall RA. Magnitude of the inflammatory response to cardiopulmonary bypass and its relation to adverse clinical outcomes. Inflamm Res. 2002 Dec;51(12):579-86. doi: 10.1007/pl00012432. PMID 12558191
- [Background] Siddiqi N, Stockdale R, Britton AM, Holmes J. Interventions for preventing delirium in hospitalised patients. Cochrane Database Syst Rev. 2007 Apr 18;(2):CD005563. doi: 10.1002/14651858.CD005563.pub2. PMID 17443600
- [Background] Jorden VSB, et al. Dexmedetomidine: clinical update. Semin Anesth Periop Med Pain 2002;21:265-74.
- [Background] Iirola T, Aantaa R, Laitio R, Kentala E, Lahtinen M, Wighton A, Garratt C, Ahtola-Satila T, Olkkola KT. Pharmacokinetics of prolonged infusion of high-dose dexmedetomidine in critically ill patients. Crit Care. 2011;15(5):R257. doi: 10.1186/cc10518. Epub 2011 Oct 26. PMID 22030215
- [Background] Liu C, Zhang Y, She S, Xu L, Ruan X. A randomised controlled trial of dexmedetomidine for suspension laryngoscopy. Anaesthesia. 2013 Jan;68(1):60-6. doi: 10.1111/j.1365-2044.2012.07331.x. Epub 2012 Oct 29. PMID 23106186
- [Background] Gozalo-Marcilla M, Hopster K, Gasthuys F, Hatz L, Krajewski AE, Schauvliege S. Effects of a constant-rate infusion of dexmedetomidine on the minimal alveolar concentration of sevoflurane in ponies. Equine Vet J. 2013 Mar;45(2):204-8. doi: 10.1111/j.2042-3306.2012.00613.x. Epub 2012 Aug 1. PMID 22853551
- [Background] Bekker A, Haile M, Kline R, Didehvar S, Babu R, Martiniuk F, Urban M. The effect of intraoperative infusion of dexmedetomidine on the quality of recovery after major spinal surgery. J Neurosurg Anesthesiol. 2013 Jan;25(1):16-24. doi: 10.1097/ANA.0b013e31826318af. PMID 22824921
- [Background] Shim JJ, Leung JM. An update on delirium in the postoperative setting: prevention, diagnosis and management. Best Pract Res Clin Anaesthesiol. 2012 Sep;26(3):327-43. doi: 10.1016/j.bpa.2012.08.003. PMID 23040284
- [Background] Park JK, Cheong SH, Lee KM, Lim SH, Lee JH, Cho K, Kim MH, Kim HT. Does dexmedetomidine reduce postoperative pain after laparoscopic cholecystectomy with multimodal analgesia? Korean J Anesthesiol. 2012 Nov;63(5):436-40. doi: 10.4097/kjae.2012.63.5.436. Epub 2012 Nov 16. PMID 23198038
- [Background] Anger KE. Dexmedetomidine: a review of its use for the management of pain, agitation, and delirium in the intensive care unit. Curr Pharm Des. 2013;19(22):4003-13. doi: 10.2174/1381612811319220009. PMID 23228319
- [Background] Oto J, Yamamoto K, Koike S, Onodera M, Imanaka H, Nishimura M. Sleep quality of mechanically ventilated patients sedated with dexmedetomidine. Intensive Care Med. 2012 Dec;38(12):1982-9. doi: 10.1007/s00134-012-2685-y. Epub 2012 Sep 8. PMID 22961436
- [Background] Oto J, Yamamoto K, Koike S, Imanaka H, Nishimura M. Effect of daily sedative interruption on sleep stages of mechanically ventilated patients receiving midazolam by infusion. Anaesth Intensive Care. 2011 May;39(3):392-400. doi: 10.1177/0310057X1103900309. PMID 21675058